CLINICAL TRIAL: NCT06320223
Title: PROMISE Registry on Standardized Evaluation of PSMA-PET and Outcome in Prostate Cancer
Brief Title: PROMISE PET Registry on PSMA-PET and Outcome in Prostate Cancer
Acronym: PROMISE-PET
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Sponsor
Other Study IDs: PROMISE PET Registry
Record Dates: First submitted 2024-03-06; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Prostate Cancer; PET/CT; Survivorship; PSMA
Keywords: Prostate Cancer; PET/CT; Survivorship; PSMA; Nuclear Medicine; Imaging; Oncology; Urology
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prostate cancer patients with PSMA PET: Inclusion:
  * Adult patients with
  * biopsy/histo proven prostate cancer who
  * underwent PSMA PET (any type)
  * for staging or re-staging at any stage and who
  * have at least 3-year overall survival follow-up data available will be included consecutively.
  Exclusion:
  * Patients with neuroendocrine prostate cancer
  * Patients with metastasized or disseminated malignancy other than prostate cancer.

SUMMARY:
Background:

PROMISE criteria have been defined for standardized reporting of Prostate-Specific Membrane Antigen (PSMA) PET whole-body stage of prostate cancer. PSMA PET disease extent by PROMISE has been associated with oncologic outcome.

Need:

Improved prognostication across various stages of prostate cancer is needed for management guidance and study design.

Aim:

1. To assess the prognostic value of PSMA PET
2. To compare the prognostic value of PSMA PET with clinical prognostic scores in patients with prostate cancer at various disease stages

Inclusion:

* Adult patients with
* biopsy/histo proven prostate cancer who
* underwent PSMA PET (any type)
* for staging or re-staging at any stage and who
* have at least 3-year overall survival follow-up data available will be included consecutively.

Exclusion:

* Patients with neuroendocrine prostate cancer
* Patients with metastasized or disseminated malignancy other than prostate cancer

DETAILED DESCRIPTION:
Background:

Prostate Cancer Molecular Imaging Standardized Evaluation (PROMISE) criteria have been defined for standardized reporting of Prostate-Specific Membrane Antigen (PSMA) Positron-Emission-Tomography (PET) whole-body stage of prostate cancer [Seifert et al. European Urology 2023]. PSMA PET disease extent by PROMISE has been associated with relevant oncologic outcome, specifically overall survival in patients with various stages of prostate cancer.

Need:

Improved risk assessment across various stages of prostate cancer is urgently needed for guidance of clinical management and prospective study design.

Aim:

1. To assess the prognostic value of PSMA PET, summarized by PROMISE [Seifert et al EurUrol23]
2. To compare the prognostic value of PSMA PET with established clinical prognostic scores in patients with prostate cancer at various disease stages
3. To assess the association of PSMA PET stage with management, laboratory findings, histopathology findings or patient characteristics

Eligibility:

Adult patients with biopsy/histo proven prostate cancer who underwent PSMA PET for staging at various stages will be included consecutively. All stages will be included: Primary (Initial Staging), BCR (Biochemical Recurrence), nmCRPC (conventional non-metastatic castration-resistant prostate cancer), mHSPC (conventional metastatic hormone-sensitive prostate cancer), mCRPC (conventional metastatic castration-resistant prostate cancer) and advanced mCRPC.

Inclusion:

* Adult patients with
* histopathology proven prostate cancer who
* underwent PSMA PET (any type)
* for staging or re-staging at any stage and who
* have at least 3-year overall survival follow-up data available will be included consecutively.

Exclusion:

* Patients with neuroendocrine prostate cancer
* Patients with metastasized or disseminated malignancy other than prostate cancer

Statistical considerations:

This is an open registry study. The more data sets are contributed, the more precisely the diagnostic accuracy and prognostic value of PSMA PET can be determined for the overall cohort and subgroups.

Prognostic value of variables from PSMA-PET (PROMISE parameters, PSMA-Volume, Standardized Uptake Value (SUV) among other) and patient characteristics will be assessed by regression analysis and correlation analysis. Hazard ratio (95% Confidence Interval) and Concordance Index for the prediction of primary and secondary endpoints will be calculated. Primary endpoint is the association with overall survival. Secondary endpoints are the association with progression-free survival, management and other characteristics.

Central Database:

Data will be stored centrally in a RedCap Database with 3-step authentication at the sponsor site.

Recurring Data Entry:

Data entry will be conducted repeatedly at about 3 to 6 month intervals.

ELIGIBILITY:
Inclusion:

* Adult patients with
* biopsy/histo proven prostate cancer who
* underwent PSMA PET (any type)
* for staging or re-staging at any stage and who
* have at least 3-year overall survival follow-up data available will be included consecutively.

Exclusion:

* Patients with neuroendocrine prostate cancer
* Patients with metastasized or disseminated malignancy other than prostate cancer.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Study Population: Adult patients with biopsy/histo proven prostate cancer who underwent PSMA PET for staging at various stages will be included consecutively. All stages will be included: Primary, BCR, nmCRPC, mHSPC, mCRPC and advanced mCRPC.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2034-03-05 (Estimated); Study Completion 2035-03-05 (Estimated)

PRIMARY OUTCOMES:
Overall survival | up to 10 years
  Time from PSMA-PET until death

SECONDARY OUTCOMES:
Metastasis-free survival | up to 10 years
  Time from PSMA-PET until development of new metastasis on any imaging

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang P Fendler, M.D., Principal Investigator — University Hospital, Essen
Locations (1):
- University Hospital Essen, Essen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karpinski MJ, Hoberuck S, Fendler WP, Civan C, Bundschuh RA, Thomas C, Bjartell A, Tragardh E, Soeterik TFW, Evangelista L, Vondrak A, Rasul S, Forner L, Giorgio AD, Scholtissek H, Miksch J, Holzgreve A, Lanfranchi F, Rahbar K, Hofman MS, Rauscher I, Guven O, Eiber M, Ayati N, Umutlu L, Herrmann K, Hadaschik B, Emmett L. Association Between the PRIMARY Score at Staging Prostate-specific Membrane Antigen Positron Emission Tomography and Overall Survival Among Patients with Newly Diagnosed Prostate Cancer: Findings from the International, Multicenter PROMISE Registry. Eur Urol. 2025 Oct 29:S0302-2838(25)04773-6. doi: 10.1016/j.eururo.2025.10.013. Online ahead of print. PMID 41168067
- [Derived] Karpinski MJ, Husing J, Claassen K, Moller L, Kajuter H, Oesterling F, Grunwald V, Umutlu L, Kleesiek J, Telli T, Merkel-Jens A, Husing A, Kesch C, Herrmann K, Eiber M, Hoberuck S, Meyer PT, Kind F, Rahbar K, Schafers M, Stang A, Hadaschik BA, Fendler WP. Combining PSMA-PET and PROMISE to re-define disease stage and risk in patients with prostate cancer: a multicentre retrospective study. Lancet Oncol. 2024 Sep;25(9):1188-1201. doi: 10.1016/S1470-2045(24)00326-7. Epub 2024 Jul 29. PMID 39089299